CLINICAL TRIAL: NCT05803382
Title: Phase I Trial of ZEN003694 (ZEN-3694) in Combination With Capecitabine in Patients With Solid Tumors
Brief Title: Testing the Addition of an Anti-Cancer Drug, ZEN003694, to the Usual Chemotherapy Treatment (Capecitabine) for Metastatic or Unresectable Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-02652; NCI-2023-02652 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCC 23-096; 10579 (Other: UPMC Hillman Cancer Center LAO); 10579 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2023-04-06; First posted 2023-04-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Carcinoma; Metastatic Malignant Solid Neoplasm; Stage IV Colorectal Cancer AJCC v8; Unresectable Colorectal Carcinoma; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Capecitabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ZEN003694, capecitabine) (Experimental): Patients receive ZEN003694 PO QD and capecitabine PO BID 2 weeks on, 1 week off during each treatment cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI, PET/CT, and collection of blood samples throughout the trial. Patients may also undergo biopsies during screening and while on the study.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Capecitabine; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Procedure: Computed Tomography — Undergo CT and PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of ZEN003694 in combination with the usual treatment with capecitabine in treating patients with cancer that has spread from where it first started (primary site) to other places in the body (metastatic) or cannot be removed by surgery (unresectable) and that it has progressed on previous standard treatment. ZEN003694 is an inhibitor of a family of proteins called the bromodomain and extra-terminal (BET). It may prevent the growth of tumor cells that over produce BET protein. Capecitabine is in a class of medications called antimetabolites. It is taken up by cancer cells and breaks down into fluorouracil, a substance that kills cancer cells. Giving ZEN003694 in combination with capecitabine may be safe in treating patients with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability, maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of BET bromodomain inhibitor ZEN-3694 (ZEN003694 [ZEN-3694]) in combination with capecitabine in patients with solid tumors.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity of ZEN003694 (ZEN-3694) in combination with capecitabine.

II. To determine the pharmacokinetics (PK) of ZEN003694 (ZEN-3694) in combination with capecitabine.

III. To determine the pharmacodynamics (PD) of ZEN003694 (ZEN-3694) in combination with capecitabine (death receptor 5 [DR5] dynamics and apoptosis).

IV. To identify molecular subpopulations particularly sensitized to bromodomain and extra-terminal motif inhibitor (BETi) and capecitabine.

OUTLINE: This is a dose-escalation study of ZEN003694 and capecitabine, followed by a dose-expansion study.

Patients receive ZEN003694 orally (PO) once daily (QD) and capecitabine PO twice daily (BID) 2 weeks on, 1 week off during each treatment cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI), positron emission tomography (PET)/CT, and collection of blood samples throughout the trial. Patients may also undergo biopsies during screening and while on the study.

After completion of study treatment, patients are followed up for safety 30 days after the last dose, and then every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation additional criteria: Patients must have histologically confirmed cancer that is metastatic or unresectable and must have progressed on standard therapies which would have included fluorouracil (5-FU) or capecitabine
* Dose Escalation additional criteria specifically for colorectal cancer (CRC) patients: Willingness and ability to undergo a pre-treatment biopsy
* Dose Expansion additional criteria: Patients must have histologically confirmed CRC that is metastatic or unresectable and must have progressed on standard therapies which would have included 5-FU or capecitabine
* Dose Expansion additional criteria: Willingness and ability to undergo pre- and on- treatment biopsies
* Patients must have measurable disease
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of ZEN003694 (ZEN-3694) in combination with capecitabine in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Karnofsky >= 60%)
* Availability of archival tumor tissue at the time of patient enrollment for molecular profiling studies
* Prior to study dosing, previous systemic therapy must have been completed for at least five half-lives or 2 weeks, whichever is shorter
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients should be New York Heart Association Functional Classification of class 2B or better
* The effects of ZEN003694 (ZEN-3694) and capecitabine on the developing human fetus are unknown. For this reason and because BET inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women of child-bearing potential and men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of ZEN003694 (ZEN-3694) and capecitabine administration
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Previous treatment with BET inhibitors
* History of inability to tolerate capecitabine at the projected treatment dose on this trial
* Use of oral Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed
* Treatment for HIV, hepatitis B or hepatitis C only if this interferes with the current treatment (e.g. through drug-drug interactions)
* Gastrointestinal pathology or history that adversely impacts the ability to take or absorb oral medication
* Hepatic tumor burden > 30% or peritoneal carcinomatosis
* Untreated/uncontrolled central nervous system (CNS) disease
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Severe intercurrent illness or comorbidity
* Inability to comply with the protocol and/or not willing or who will not be available for follow-up assessments
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and neuropathy up to and including grade 2
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZEN003694 (ZEN-3694) or other agents used in study
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Strong inhibitors of CYP3A4 must be discontinued at least 7 days, and inducers 14 days prior to the first dose of ZEN003694 and capecitabine. Substrates of CYP1A2 with narrow therapeutic window must be avoided while taking ZEN003694
* Pregnant women are excluded from this study because ZEN003694 (ZEN-3694) is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ZEN003694 (ZEN-3694), breastfeeding should be discontinued if the mother is treated with ZEN003694 (ZEN-3694). These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose
  Adverse events and serious adverse events will be tabulated for each dose levels. As per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, the term toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Maximum tolerated dose (MTD) | During the first cycle of therapy (Cycles = 21 days)
  Defined as the highest dose level with no more than 1/6 dose-limiting toxicity.
Recommended phase 2 dose (RP2D) | Up to 30 days after last dose
  Will be determined based on the MTD and later cycle adverse event (AE) rates.

SECONDARY OUTCOMES:
Anti-tumor activity of ZEN003694 (ZEN-3694) in combination with capecitabine | Up to 12 months
  Treatment response will be assessed for all patients based on Response Evaluation Criteria in Solid Tumors version 1.1: complete response (CR), partial response (PR), stable disease (SD), and progression of disease (PD). Clinical benefit rate is defined as the addition of CR, PR and SD.
Progression free survival (PFS) | Up to 12 months
  PFS will be estimated by the Kaplan-Meier method, along with 95% confidence regions.
Objective response rate (ORR) | Up to 12 months
  Defined as the addition of CR and PR. The probability of ORR and clinical benefit rate will be estimated with exact 95% binomial confidence intervals.
Pharmacokinetics (PK) of ZEN003694 (ZEN-3694) in combination with capecitabine | Up to 12 months
  Will determine the PK of ZEN003694 (ZEN-3694) in combination with capecitabine. Capecitabine PK will be evaluated in the absence and presence of ZEN003694 (ZEN-3694) and Cmax and area under curve (AUC) will be compared with a paired test. ZEN003694 (ZEN-3694) PK will be evaluated in the presence of capecitabine and Cmax and AUC will be compared descriptively with historical data.
Pharmacodynamics (PD) of ZEN003694 (ZEN-3694) in combination with capecitabine | Up to 12 months
  Will determine PD of ZEN003694 (ZEN-3694) in combination with capecitabine. Ribonucleic acid sequencing of death receptor 5 (DR5). DR5 is expected to be increased by the combination ZEN003694 (ZEN-3694) in combination with capecitabine. Pre-post comparisons will be made within patients enrolled on the expansion cohort using a non-parametric paired test, at a significance level (alpha) of 0.05. Apoptosis by Pharmacodynamic Assay Development and Implementation Section (PADIS) lab. Panel 3 is priority, but other panels will be evaluated with remaining lysate. Apoptosis is expected to be increased by the combination ZEN003694 (ZEN-3694) in combination with capecitabine. Pre-post comparisons will be made within patients enrolled on the expansion cohort using a non-parametric paired test, at a significance level (alpha) of 0.05.
Molecular subpopulations particularly sensitized to BETi and capecitabine | Up to 12 months
  Will identify molecular subpopulations particularly sensitized to BETi and capecitabine. Based on WES of archival tissue, we will evaluate descriptively any mutations in genes relevant to DNA damage repair, signaling and (fluoropyrimidine) metabolism, any relations with peculiar response and/or toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hsu, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (22):
- United States (22):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm